CLINICAL TRIAL: NCT01146054
Title: Phase II Multi-Institutional Study to Evaluate the Efficacy of Gemcitabine and Fractionated Stereotactic Radiotherapy for Unresectable Pancreatic Adenocarcinoma
Brief Title: Phase II Gemcitabine + Fractionated Stereotactic Radiotherapy for Unresectable Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Albert Koong, Sue and Bob McCollum Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-17073; SU-02012010-4843 (Other: Stanford University); PANC0007 (Other: OnCore)
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT and Gemzar (Experimental): Before stereotactic Body Radiotherapy (SBRT) 3-5 gold fiducials are placed by endoscopic ultrasound or CT guidance. A simulation FDG-PET/CT (Fludeoxyglucose (18F) - Positron emission tomography/Computerized tomography) scan will be used for treatment planning purposes (standard free-breathing CT and respiratory-correlated 4-D (4 dimensional) pancreatic protocol CT). Patients are treated by either respiratory gated (Trilogy, Elekta, Novalis) or by respiratory tracking (CyberKnife). SBRT is delivered in 5 fractions of 6.6 Gy by LINAC-based or CyberKnife based radiotherapy over a five-day period. Gemcitabine, cycles should resume/start up to 4 weeks following SBRT on a 3-week on, 1-week off schedule. Initial follow up is at 4, 6, 9 and 12 months and then for years 2-5 is every 3-6 months.
  Interventions: Device: CyberKnife based stereotactic radiotherapy; Drug: Gemcitabine; Drug: Fludeoxyglucose (18F) (FDG)

INTERVENTIONS:
Device: CyberKnife based stereotactic radiotherapy — 1. Initial orthogonal images will be obtained to confirm location of fiducial seeds.
  2. Synchrony respiratory tracking system must be used to correct for respiratory associated tumor motion. This system utilizes a series of optical diodes placed upon the patient's chest wall. While the orthogonal images are obtained, the computer generates a model correlating the position of the chest wall with the position of the internal fiducials. This model is continuously updated during treatment to correct for subtle changes in tumor location.
  3. Quality assurance will be performed as per standard practice at each participating institution.
  Other Names: Trilogy(Varian, Palo Alto CA); Novalis (BrainLab, Feldkirchen, Germany); Synergy (Elekta AB, Stockholm, Sweden),
Drug: Gemcitabine — Treatment calculated per the needs of each patient and given at the instruction of the investigator; iv (intravenous).
  Other Names: Gemzar
Drug: Fludeoxyglucose (18F) (FDG) — FDG-PET/CT scan is used in treatment planning. Treatment with 18F-FDG is calculated per the needs of each patient and given at the instruction of the investigator; iv
  Other Names: fluorodeoxyglucose (18F); 18F-FDG; FDG

SUMMARY:
This multi-institutional trial aims to evaluate the potential benefit and side effects of adding fractionated stereotactic body radiotherapy/surgery (SBRT) before and after chemotherapy with gemcitabine for locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Treatment on this protocol requires placement of 3-5 gold (99.9% pure, 1-5 mm length, or visicoils) fiducials for targeting purposes. The fiducials will be used as surrogates for targeting the daily tumor position during treatment. The fiducials will be placed directly into the tumor and/or periphery under endoscopic ultrasound or CT guidance. Gemcitabine prior to SBRT is optional. If given, up to 3 weeks in a 6-week period is allowable, and may be given prior to study enrollment. Administration should be on a 3-week on, 1-week off schedule, weekly at 1,000 mg/m2. Simulation should be done 5 days or more following placement of fiducials. For simulation patients will be positioned supine in an Alpha Cradle or equivalent immobilization device will be custom made for each patient. Standard free-breathing CT and respiratory-correlated 4-D pancreatic protocol CT will be obtained on each patient The 4D-CT scan will be used for characterizing target motion during quiet respiration. Following simulation, patients may be treated either in a respiratory gated (Trilogy, Elekta, Novalis) or a respiratory tracking (Cyberknife) manner. The selection of which radiotherapy treatment machine to use is left to each investigator. All patients will receive 5 fractions of 6.6 Gy delivered over a five-day period. Ideally all 5 fractions should be delivered Monday through Friday, however it may be delivered over 2 weeks as long as the patient receives at least 2 fractions a week. Gemcitabine, cycles should resume up to 4 weeks following SBRT on a 3-week on, 1-week off schedule, administered weekly at 1,000 mg/m2.A detailed medical history with physical examination and quality of life assessment will be performed at 4 months, 6 months, 9 months and 1 year. A follow-up visit at 4 weeks is optional and may be done by patient's Medical Oncologist. Scans may be done at 4-6 week visit if patient is being re-evaluated for resection.

In years 2-5 the follow up interval will be every 3-6 months, as determined by the investigator at each participating institution. Follow up intervals may also be more frequent as indicated clinically. A complete blood count (CBC), comprehensive chemistry panel, tumor marker studies, and quality of life assessment will be performed at each follow-up interval until death. As permitted by each participating institution, separate samples of blood will be drawn and retained for research efforts to develop novel serum biomarkers.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Histologically confirmed adenocarcinoma of the pancreas.

3.1.2 Unresectable disease as determined by a pancreatic cancer surgeon and assessment at a GI oncology tumor board (JHU - Johns Hopkins University, SU - Stanford University, or MSKCC - Memorial Sloan Kettering Cancer Center).

3.1.3 Up to 3 weeks of gemcitabine chemotherapy is allowed prior to SBRT.

3.1.4 Pancreatic tumors must be less than 7.5 cm in greatest axial dimension (or <1000 cc in volume) at the time of treatment planning.

3.1.5 No prior upper abdominal or liver radiation therapy.

3.1.6 No chemotherapy within 2 weeks of radiotherapy, or chemotherapy within parameters set by Investigator for each institution.

3.1.7 Age >=18 years.

3.1.8 No infections requiring systemic antibiotic treatment.

3.1.9 Karnofsky >= 70% (see Appendix III).

3.1.10 Patients must have acceptable organ and marrow function as defined below (within 1 month prior to radiotherapy):

* leukocytes: >=3,000/microliter (uL)
* absolute neutrophil count: >=1,500uL
* platelets: >=100,000/uL
* total bilirubin: within 1.5 times (1.5X) normal institutional limits
* AST (aspartate aminotransferase)(SGOT -Serum glutamic oxaloacetic transaminase)/ALT(alanine aminotransferase)(SGPT-serum glutamic-pyruvic transaminase): <=2.5 X institutional upper limit of normal
* creatinine: within normal institutional limits

OR

- creatinine clearance: >=60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal

3.1.11 The effects of radiation on the developing human fetus at recommended therapeutic doses can result in death of the fetus. If a woman is of child-bearing potential, a negative urine or serum pregnancy test must be demonstrated prior to treatment. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for up to 4 weeks following the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

3.1.12 Ability to understand and the willingness to sign a written informed consent document.

3.1.13 Life expectancy > 6 months

Exclusion Criteria:

3.2.1 Patients who have had prior radiotherapy to the upper abdomen.

3.2.2 Patients receiving more than 1 cycle of gemcitabine chemotherapy or other therapy prior to SBRT.

3.2.3 Children are excluded because pancreatic tumors rarely occur in this age group. Furthermore, treatment requires a great deal of patient cooperation including the ability to lie still for several hours in an isolated room.

3.2.4 No laboratory personnel will be included.

3.2.5 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

3.2.6 Any concurrent malignancy other than non-melanoma skin cancer, non-invasive bladder cancer, or carcinoma in situ of the cervix. Patients with a previous malignancy without evidence of disease for > 5 years will be allowed to enter the trial.

3.2.7 Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 4 weeks after the study are excluded. This applies to any woman who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months, or women on hormone replacement therapy with serum FSH (follicle stimulating hormone) levels greater than 35 IU/mL (international units/milliliter). A negative urine or serum pregnancy test must be obtained within 72 hours prior to the start of study medication in all women of childbearing potential. Male subjects must also agree to use effective contraception for the same period as above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-10; Primary Completion 2013-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Koong, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited during new patient clinical visits between 10/22/2009 - 08/14/2013 at Stanford University, Johns Hopkins University and Memorial Sloan-Kettering Cancer Center. Study details were explained by the physician and consent was obtained by the physician or study coordinator according to good clinical practices.
Groups:
- SBRT and Gemzar: 3-5 gold fiducials are placed by endoscopic ultrasound or CT guidance. A simulation FDG-PET/CT (Fludeoxyglucose 18F-positron emission tomography/computerized tomography) scan will be used for treatment planning purposes (standard free-breathing CT and respiratory-correlated 4-D (4 dimensional) pancreatic protocol CT). Patients are treated by either respiratory gated (Trilogy, Elekta, Novalis) or by respiratory tracking (CyberKnife). SBRT is delivered in 5 fractions of 6.6 Gy by LINAC-based or CyberKnife based radiotherapy over a five-day period. Gemcitabine, cycles starts within 4 weeks of SBRT on a 3-week on, 1-week off schedule. Initial follow up is at 4, 6, 9 and 12 months and then for years 2-5 is every 3-6 months.
  Fludeoxyglucose (18F): FDG-PET/CT scan is used in treatment planning. Treatment with 18F-FDG is calculated per the needs of each patient and given at the instruction of the investigator; iv
Period: Overall Study
Arm/Group | SBRT and Gemzar
Started | 59
Completed | 49
Not Completed | 10
Not completed — Did not meet dose constraints for SBRT | 5
Not completed — Rapid tumor progression | 2
Not completed — Other illness precluded treatment | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The entire cohort is analyzed.
Groups:
- SBRT and Gemzar: Before stereotactic Body Radiotherapy (SBRT) 3-5 gold fiducials are placed by endoscopic ultrasound or CT guidance. A simulation FDG-PET/CT (Fludeoxyglucose (18F)) scan will be used for treatment planning purposes (standard free-breathing CT and respiratory-correlated 4-D pancreatic protocol CT). Patients are treated by either respiratory gated (Trilogy, Elekta, Novalis) or by respiratory tracking (CyberKnife). SBRT is delivered in 5 fractions of 6.6 Gy by LINAC-based or CyberKnife based radiotherapy over a five-day period. Gemcitabine, cycles should resume/start up to 4 weeks following SBRT on a 3-week on, 1-week off schedule. Initial follow up is at 4, 6, 9 and 12 months and then for years 2-5 is every 3-6 months.
  Device: CyberKnife based stereotactic radiotherapy
Arm/Group | SBRT and Gemzar
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 33
Age, Continuous [Median (Full Range); unit: Years] | 67 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 49
Baseline Cancer Antigen 19-9 (CA19-9) [Count of Participants; unit: Participants] — Tumor marker from blood draw during routine labs.
  Participants
    CA 19-9 < 90 U/mL | 18
    CA 19-9 >= 90 U/mL | 27
Eastern Cooperative Oncology Group performance status (ECOG PS) [Count of Participants; unit: Participants] — Performance status assessed by the physician prior to treatment. ECOG 0= Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  ECOG 1 = Symptomatic but completely ambulatory ECOG 2 = Symptomatic, <50% in bed during the day ECOG 3 = Symptomatic, >50% in bed, but not bedbound ECOG 4 = Bedbound, Completely disabled. Cannot carry on any self-care. ECOG 5 = Death
  Participants
    ECOG 0 | 21
    ECOG 1 | 28
Treating Institutions [Count of Participants; unit: Participants]
  Johns Hopkins University | 32
  Memorial Sloan-Kettering Cancer Center | 3
  Stanford University | 14

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Rate of (Grade 2 or Greater) Gastrointestinal Toxicity Attributable to Gemcitabine and Fractionated SBRT at One Year.
Description: Grade 2 or greater late gastritis, fistula, enteritis, or ulcer or late grade 3-4 gastrointestinal toxicity at one year.
Time Frame: One year.
Population: The whole cohort was analyzed.
Measure: Number; unit: Number of toxicities.
Groups:
- SBRT and Gemzar: 3-5 gold fiducials are placed by endoscopic ultrasound or CT guidance. A simulation FDG-PET/CT (Fludeoxyglucose (18F)) scan will be used for treatment planning purposes (standard free-breathing CT and respiratory-correlated 4-D pancreatic protocol CT). Patients are treated by either respiratory gated (Trilogy, Elekta, Novalis) or by respiratory tracking (CyberKnife). SBRT is delivered in 5 fractions of 6.6 Gy by LINAC-based or CyberKnife based radiotherapy over a five-day period. Gemcitabine, cycles starts within 4 weeks of SBRT on a 3-week on, 1-week off schedule. Initial follow up is at 4, 6, 9 and 12 months and then for years 2-5 is every 3-6 months.
  Fludeoxyglucose (18F): FDG-PET/CT scan is used in treatment planning. Treatment with 18F-FDG is calculated per the needs of each patient and given at the instruction of the investigator; iv
Arm/Group | SBRT and Gemzar
Number analyzed (Participants) | 49
Number of toxicities. | 5

2. Secondary Outcome: Evaluate Acute Gastrointestinal Toxicity up to 3 Months of Treatment.
Description: Acute grade 2 or greater gastritis, fistula, enteritis, or ulcer or any other grade 3-4 gastrointestinal toxicity within 3 months of treatment.
Time Frame: Within 3 months of treatment.
Population: Whole cohort.
Measure: Number; unit: Number of toxicities.
Arm/Group | SBRT and Gemzar
Number analyzed (Participants) | 49
Number of toxicities. | 14

3. Secondary Outcome: To Evaluate Progression Free Survival Following Gemcitabine and SBRT for up to 5 Years of Follow up .
Description: Time to progression free survival is measured from start of SBRT treatment until first progression event or death, which ever comes first. If the patient did not have an event, then the patient was censored at the last follow up.
  The analysis was a Kaplan-Meier curve and the outcome was the median time to progression free survival.
Time Frame: Up to 5 years of follow up.
Population: The whole cohort.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SBRT and Gemzar
Number analyzed (Participants) | 49
Months | 7.8 [5.8 to 10.2]

4. Secondary Outcome: To Determine the Overall Survival in Pancreatic Cancer Patients Treated With Gemcitabine and SBRT for up to 5 Years of Follow up.
Description: Time to death was measured from start of treatment to until death. If death was not observed, the patient was censored at last follow up.
Time Frame: Up to 5 years of follow up.
Population: The entire cohort.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SBRT and Gemzar
Number analyzed (Participants) | 49
Months | 13.9 [10.2 to 16.7]

5. Secondary Outcome: Proportion of Participants Achieving Freedom From Local Progression (FFLP) in Patients Treated With Gemcitabine Followed by Fractionated Stereotactic Body Radiotherapy (SBRT) for up to 5 Years of Follow up.
Description: Freedom from local progression is defined as the time from start of SBRT treatment to local progression, with death as a competing risk. If the patient neither died nor experienced local progression, then patient was censored at last follow up.
  The data was analyzed in a competing risk model and the outcome reported was the 1 year cumulative incidence rate.
Time Frame: Up to 5 years of follow up.
Measure: Number (95% Confidence Interval); unit: Proportion of participants with FFLP
Arm/Group | SBRT and Gemzar
Number analyzed (Participants) | 49
Proportion of participants with FFLP | 0.78 [0.60 to 0.89]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment to end of follow up (5 years).
Arm/Group | SBRT and Gemzar
Serious Adverse Events (participants affected / at risk) | 6/49
Other Adverse Events (participants affected / at risk) | 25/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT and Gemzar (N=49)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) — Grade 4 duodenal ulcer 43 days after completion of SBRT.
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Subject died of dehydration secondary to C. Difficile infection.
Sepsis (Infections and infestations) | 1 (1) — During a stent change for cholangitis, the bile duct was perforated leading to Klebsiella pneumoniae sepsis, from which the patient died.
Duodenal Fistula (Gastrointestinal disorders) | 1 (1) — Grade 4 fistula between the tumor and the duodenum. Patient discharged to hospice and died 2 weeks later.
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) — Grade 3 duodenal hemorrhage secondary to stent migration.
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) — Grade 5 GI bleed due to direct tumor extension into the duodenum resulting in death.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT and Gemzar (N=49)
Abdominal Pain (Gastrointestinal disorders) | 12 (12)
Anorexia (Metabolism and nutrition disorders) | 13 (13)
Constipation (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 14 (14)
Lymphocyte count decreased (Investigations) | 14 (14)
Platelet Count Decreased (Investigations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No